CLINICAL TRIAL: NCT04208529
Title: A Long-term Follow-up Study of Subjects With β-thalassemia or Sickle Cell Disease Treated With Autologous CRISPR-Cas9 Modified Hematopoietic Stem Cells (CTX001)
Brief Title: A Long-term Follow-up Study in Participants Who Received CTX001
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VX18-CTX001-131; 2024-512654-19-00 (Other: EU CT Number)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-08

CONDITIONS: Beta-Thalassemia; Thalassemia; Sickle Cell Disease; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Sickle Cell Anemia
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn | interventions — exagamglogene autotemcel

STUDY DESIGN:
Intervention Model Description: Long Term Safety Follow-up
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CTX001 (Experimental): All participants who complete or discontinue one of the multiple parent studies (CTX001-111, CTX001-121, CTX001-141, CTX001-151, CTX001-161 and CTX001-171) after CTX001 infusion will be asked to participate in this long-term follow-up study.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — CTX001 infusion.
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a multi-site, open- label rollover study to evaluate the long-term safety and efficacy of CTX001 in pediatric and adult participants who received CTX001 in parent studies 111 (NCT03655678) 141 (NCT05356195) or 161 (NCT05477563) (transfusion-dependent β-thalassemia [TDT] studies) or Study 121 (NCT03745287) or 151 (NCT05329649), 161(NCT05477563),171 (NCT05951205) (severe sickle cell disease [SCD] studies).

ELIGIBILITY:
Inclusion Criteria:

* Participants (or his or her legally appointed and authorized representative or guardian) must sign and date informed consent form (ICF) and, where applicable, an assent form
* Participants must have received CTX001 infusion in a parent study

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2039-09-30 (Estimated); Study Completion 2039-09-30 (Estimated)

PRIMARY OUTCOMES:
New malignancies | Signing of informed consent up to 15 years post CTX001 infusion
New or worsening hematologic disorders | Signing of informed consent up to 15 years post CTX001 infusion
All-cause mortality | Signing of informed consent up to 15 years post CTX001 infusion
Serious adverse events (SAEs) | Signing of informed consent up to 15 years post CTX001 infusion
CTX001-related adverse events (AEs) | Signing of informed consent up to 15 years post CTX001 infusion

SECONDARY OUTCOMES:
TDT and SCD: Total Hemoglobin (Hb) concentration over time | Up to 15 years post CTX001 infusion
TDT and SCD: Fetal Hemoglobin (HbF) concentration over time | Up to 15 years post CTX001 infusion
TDT and SCD: Proportion of alleles with intended genetic modification present in peripheral blood over time | Up to 15 years post CTX001 infusion
TDT and SCD: Proportion of alleles with intended genetic modification present in CD34+ cells of the bone marrow over time | Up to 15 years post CTX001 infusion
TDT and SCD: Change in patient-reported outcome (PRO) over time in participants ≥18 years of age assessed using EuroQol quality of life scale (EQ-5D-5L) for participants from study 111,121 and 171 only | Up to 5 years post CTX001 infusion
TDT and SCD: Change in PROs over time in participants ≥18 years of age assessed using functional assessment of cancer therapy-bone marrow transplant (FACT-BMT) questionnaire for participants from study 111, 121, 161 and 171 only | Up to 5 years post CTX001 infusion
TDT and SCD: Change in PROs over time in participants <18 years assessed using EQ-5D-Youth (EQ-5D-Y) from study 111,121,141,151 and 171 only | Up to 5 years post CTX001 infusion
TDT and SCD: Change in PROs over time in participants <18 years assessed using pediatric quality of life inventory (PedsQL) Core | Up to 5 years post CTX001 infusion
TDT: Proportion of participants achieving transfusion independence for at least 12 consecutive months (TI12) | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
TDT: Proportion of participants achieving transfusion independence for at least 6 consecutive months (TI6) | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
TDT: Proportion of participants achieving at least 95%, 90%, 85%, 75%, 50% reduction from baseline in annualized volume of RBC transfusions starting after month 10 after CTX001 infusion for participants who have not achieved TI12 | From Month 10 up to 15 years post-CTX001 infusion
TDT: Duration of transfusion free in participants who have achieved TI12 | From 60 days after last RBC transfusion up to 15 years post CTX001 infusion
TDT: Relative reduction from baseline in annualized volume of RBC transfusions starting after Month 10 after CTX001 infusion for participants who have not achieved TI12 | From Month 10 up to 15 years post-CTX001 infusion
TDT: Iron overload as measured by liver iron concentration (LIC), cardiac iron concentration (CIC), and ferritin for beta-Thalassemia participants | Up to 8 years post CTX001 infusion for LIC; up to 5 years post CTX001 infusion for CIC and up to 15 years post CTX001 infusion for ferritin
TDT: Proportion of participants receiving iron removal therapy over time | Up to 15 years post CTX001 infusion
SCD: Proportion of participants who have not experienced any severe vaso-occlusive crises (VOC) for at least 12 consecutive months (VF12) | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Proportion of participants with SCD free from inpatient hospitalization for severe VOCs sustained for at least 12 months (HF12) | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Proportion of participants with at least 90 percent (%), 80%, 75% or 50% reduction in annualized rate of severe VOCs | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Relative change from baseline in annualized rate of severe VOCs | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Duration of severe VOC free in participants who have achieved VF12 | From 60 days after last RBC transfusion up to 15 years post CTX001 infusion
SCD: Relative change from baseline in rate of inpatient hospitalizations for severe VOCs | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Relative change from baseline in annualized duration of hospitalization for severe VOCs | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Proportion of participants with sustained HbF ≥20% for at least 3 months | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Proportion of participants with sustained HbF ≥20% for at least 6 months | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Proportion of participants with sustained HbF ≥20% for at least 12 months | From 60 days after last RBC transfusion up to 15 years post-CTX001 infusion
SCD: Change in volume of RBCs transfused for SCD-related indications over time | Up to 15 years post CTX001 infusion
SCD: Change from baseline in reticulocytes/erythrocytes over time | From baseline up to 15 years post CTX001 infusion
SCD: Change from baseline in lactate dehydrogenase (LDH) over time | From baseline up to 15 years post CTX001 infusion
SCD: Change from baseline in haptoglobin over time | From baseline up to 15 years post CTX001 infusion
SCD: Change from baseline in total bilirubin over time | From baseline up to 15 years post CTX001 infusion
SCD: Change from baseline in indirect bilirubin over time | From baseline up to 15 years post CTX001 infusion
SCD: Change in SCD-specific PROs over time in participants ≥18 years of age assessed using adult sickle cell quality of life measurement system (ASCQ-Me) (participants from Study 121,161 and 171 only) | Up to 5 years post CTX001 infusion
SCD: Change in SCD-specific PROs over time in participants <18 years of age assessed using PedsQL Generic Core SCD module from studies 111,121,141,151,161 and 171 | Up to 5 years post CTX001 infusion
SCD: Change in PRO over time assessed using 11-point numerical rating scale (NRS) | Up to 5 years post CTX001 infusion
SCD: Change in PROs over time assessed using Wong Baker FACES pain scale | Up to 5 years post CTX001 infusion
SCD: Change in PROs over time using face, legs, activity, cry, consolability (FLACC) behavioral pain scale | Up to 5 years post CTX001 infusion

CONTACTS AND LOCATIONS:
Locations (19):
- United States (9):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago - Hematology, Chicago, Illinois
  - Herbert Irving Pavilion - Hematology, New York, New York
  - New York Presbyterian Hospital - Morgan Stanley Children's Hospital, New York, New York
  - Levine Children's Hospital - Hematology, Charlotte, North Carolina
  - The Children's Hospital of Philadelphia - Hematology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - TriStar Medical Group Children's Specialists - Pediatric Oncology, Nashville, Tennessee
  - Methodist Healthcare System of San Antonio, Methodist Hospital, Methodist Children's Hospital, San Antonio, Texas
- Hopital Universitaire des Enfants Reine Fabiola (HUDERF) - Hematology, Brussels, Belgium
- Canada (3):
  - Hospital for Sick Children - Hematology, Toronto
  - Toronto General Hospital - Hematology, Toronto
  - St. Paul's Hospital - Hematology, Vancouver
- Germany (3):
  - University Hospital Duesseldorf - Department of Pediatric Oncology, Hematology and Clinical Immunology, Düsseldorf
  - Center for Pediatric Clinical Studies (CPCS), Klinik Für Kinder- Und Jugendmedizin
  - Regensburg University Hospital, Clinic and Polyclinic for Paediatric and Adolescent Medicine, Regensburg
- IRCSS Ospedale Pediatrico Bambino Gesu - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica, Rome, Italy
- United Kingdom (2):
  - Hammersmith Hospital - Haematology Dept, London
  - University College London Hospital NHS Foundation - Main, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Fuente J, Frangoul H, Lang P, Wall D, Meisel R, Corbacioglu S, Li AM, Shah AJ, Carpenter B, Kwiatkowski JL, Mapara MY, Liem RI, Rupprecht J, Kuo KHM, Merkeley H, Algeri M, Smith W, Kohli P, Li N, Rubin J, Zhang S, Hobbs W, Locatelli F. Improvements in health-related quality of life in patients with transfusion-dependent beta-thalassemia after exagamglogene autotemcel. Blood Adv. 2025 Dec 23;9(24):6502-6510. doi: 10.1182/bloodadvances.2025016702. PMID 40862696
- [Derived] Sharma A, Locatelli F, Bhatia M, Molinari L, Mapara MY, Liem RI, Dedeken L, Wall D, Eckrich MJ, Kuo KHM, Smith W, Imren S, Kohli P, Li N, Liu T, Rubin J, Hobbs W, Grupp SA, Frangoul H. Improvements in health-related quality of life in patients with severe sickle cell disease after exagamglogene autotemcel. Blood Adv. 2025 Dec 23;9(24):6481-6490. doi: 10.1182/bloodadvances.2025016701. PMID 40857358